CLINICAL TRIAL: NCT04511065
Title: Impact of the Use of a Computer-based Newsletter, Using a Virtual Delivery of Intervention, on Literacy Engagement and Reading Achievement of Middle School-aged Students
Brief Title: Computer Based Newsletter and Literacy Engagement of Middle-school Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Turquessa Francis, Clinical Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004610
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Reading Problem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be provided with a survey to determine areas of interest to guide the 7-week literacy intervention plan of completing a newsletter. Students will complete the newsletter virtually using secure Zoom meetings 2x per week for 30 minutes per session. The results of the GORT 5 and TOC will be used to determine the baseline reading skills of the students and each researcher will use the results of the assessments to guide the intervention with the newsletter topic that is chosen by the student. For example, if the GORT 5 notes deficiency with reading accuracy, the focus of the intervention will be ensuring that reading accuracy is a focus of the summary that is crafted by the student for the newsletter.
  Interventions: Other: Newsletter using a virtual mode of delivery
- Control Group (No Intervention): The control group will not participate in the newsletter creation for the 7-week study period. These students will engage in the after-school programs at the Center, some of which may be literacy-based, but not the prescriptive model that is being followed by the researchers.

INTERVENTIONS:
Other: Newsletter using a virtual mode of delivery — Newsletter creation where topics in the newsletter are chosen by participants in the intervention group.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to improve motivation for reading by implementing a computer-based newsletter and examine the effects on the literacy engagement and reading achievement of middle school-aged students. Research questions to be answered: 1. Does the provision of a computer-based newsletter intervention improve literacy engagement on middle school students in comparison to their pretest scores? 2. Does the provision of computer-based newsletter intervention improve the reading achievement of middle school students in comparison to their pretest scores?

DETAILED DESCRIPTION:
For children where consent was provided by a parent or legal guardian, an assent form will be completed by the child for the child to also consent to participate in the study. Once consent and assent have been received, the student's reading skills will be assessed using the Gray Oral Reading Test 5 (GORT 5) and Test of Orthographic Competence (TOC). The student will also be assessed using a modified Inventory of Reading Occupations (IRO) to determine their access to reading materials and their perceived proficiency with the reading tasks. From the results of the GORT 5 and TOC, inclusion criteria will be used to determine if students will be included in the study. Once the inclusion criteria have been determined for all students, students will be randomly placed in either a control or intervention group.

The intervention group will be provided with a survey to determine areas of interest to guide the 7-week literacy intervention plan of completing a newsletter. Students will complete the newsletter virtually using secure Zoom meetings 2x per week for 30 minutes per session. The results of the Gray Oral Reading Tets 5 (GORT 5) and Test of Orthographic Competence (TOC) will be used to determine the baseline reading skills of the students and each researcher will use the results of the assessments to guide the intervention with the newsletter topic that is chosen by the student. For example, if the GORT 5 notes a deficiency in reading accuracy, the focus of the intervention will be ensuring that reading accuracy is a focus of the summary that is crafted by the student for the newsletter.

At the end of 7-weeks, the control group and intervention group will be re-administered the Gray Oral Reading Test 5 and Test of Orthographic Competence to determine reading skills. Students will also be provided with the modified Inventory of Reading Occupations (IRO). The control and intervention group's GORT 5, TOC, and modified IRO scores will be analyzed to find out the differences between the groups in reading skills (using the GORT 5 and TOC) and reading interest/perceived reading proficiency (using the modified IRO).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be in After-school participants ages 10-13 years old and in grades 6-8.
2. Have access to a computer: laptop, Chromebook, or desktop.
3. Can identify and press all keys on a keyboard.
4. Can use a mouse to navigate on a computer.
5. Have internet access at home or center.
6. Computer system has the capability to download Zoom.
7. One grade equivalent or more below in areas of: fluency, rate, accuracy, or comprehension on Gray Oral Reading Test 5 (GORT 5).
8. Standard score in the below average range on the Test of Orthographic Competence (TOC).
9. Participants must speak, read, and write in English

Exclusion Criteria:

- 1. Students who do not have access to a computer, internet, and Zoom access at home.

2. Students who do not speak, read, and write in English.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Reading Skills of Middle-School Aged Children | These assessments will be administered at the start of the study and at the end of the study. Total timeframe from Time 1 to Time 2 is 7 weeks.
  Reading skills will be assessed using the Gray Oral Reading Test 5 (GORT 5) and the Test of Orthographic Competency (TOC). The Gray Oral Reading Test 5 assesses oral reading skills of individuals ages 6-23 years old, in the areas of rate, accuracy, fluency, and comprehension. The Test of Orthographic Competence assesses reading skills of children ages 6-17 years old, looking at proficiency with letters, spelling, punctuation, abbreviations and special symbols.

SECONDARY OUTCOMES:
Literacy Engagement of Middle-School Aged Children | This assessment will be administered at the start of the study and at the end of the study. Total timeframe from Time 1 to Time 2 is 7 weeks.
  The researchers will also administer the modified Inventory of Reading Occupations (modified-IRO), a literacy engagement scale created by the investigators using the two standardized assessments, Inventory of Reading Occupations Pediatric version, and Inventory of Reading Occupations Adult version.

CONTACTS AND LOCATIONS:
Overall Officials: Turquessa Francis, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Grajo LC, Candler C, Bowyer P, Schultz S, Thomson J, Fong K. Determining the Internal Validity of the Inventory of Reading Occupations: An Assessment Tool of Children's Reading Participation. Am J Occup Ther. 2016 May-Jun;70(3):7003220010p1-9. doi: 10.5014/ajot.2016.017582. PMID 27089292
- [Background] Kim, A.-H., Vaughn, S., Klingner, J. K., Woodruff, A. L., Reutebuch, C. K., & Kouzekanani, K. (2006). Improving the reading comprehension of middle school students with disabilities through computer-assisted collaborative strategic reading. Remedial and Special Education, 27(4), 235-249. doi: 10.1177/07419325060270040401